CLINICAL TRIAL: NCT01597778
Title: A Multi-Center, Phase III, Randomized Trial of RIC and Transplantation of (dUCB) Versus HLA-Haplo Related Bone Marrow for Patients With Hematologic Malignancies.(BMT CTN #1101)
Brief Title: Double Cord Versus Haploidentical (BMT CTN 1101)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN1101; 2U10HL069294-11 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Acute Lymphocytic Leukemia; Acute Myelogenous Leukemia; Burkitt's Lymphoma; Follicular Lymphoma; Hodgkin Lymphoma; Mantle Cell Lymphoma; Non-Hodgkin Lymphoma
Keywords: Haplo identical transplant; Cord blood transplant; Reduced intensity conditioning regimen; Lymphoma; Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Follicular; Hodgkin Disease; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Haploidentical Bone Marrow Transplant (Experimental): Participants will receive haploidentical bone marrow transplant using a reduced intensity conditioning regimen.
  Interventions: Biological: Haploidentical Bone Marrow Transplant
- Double Umbilical Cord Blood Transplant (Experimental): Participants will receive a double umbilical cord blood transplant using a reduced intensity conditioning regimen.
  Interventions: Biological: Double Umbilical Cord Blood Transplant

INTERVENTIONS:
Biological: Haploidentical Bone Marrow Transplant — The conditioning regimen consists of:
  Fludarabine (Flu)30 mg/m2 IV Days -6, -5, -4, -3, -2 Cyclophosphamide (Cy) 14.5 mg/kg IV Days -6, -5 Total body irradiation (TBI) 200cGy Day -1
  The GVHD prophylaxis regimen consists of:
  Cy 50 mg/kg IV Days 3, 4 Tacrolimus (IV or PO) beginning Day 5 Mycophenolate mofetil (MMF) 15 mg/kg po three times a day, maximum dose 1 g po TID beginning Day 5 until Day 35
  Arms: Haploidentical Bone Marrow Transplant
Biological: Double Umbilical Cord Blood Transplant — The preparative regimen consists of:
  Fludarabine 40 mg/m2 IV Days -6, -5, -4,-3, -2 Cyclophosphamide 50 mg/kg IV Day -6 Total Body Irradiation (TBI) 200 cGy Day -1 for patients who have received cytotoxic chemotherapy within the 3 months of enrollment or an autologous transplant within 24 months of enrollment or 300 cGy Day -1 for patients who have not received cytotoxic chemotherapy within the 3 months of enrollment and who have not received an autologous transplant within 24 months of enrollment.
  The GVHD prophylaxis regimen consists of:
  Cyclosporine beginning Day -3 with dose adjusted to maintain a trough level of 200-400 ng/mL.
  Mycophenolate mofetil (MMF) 15 mg/kg po three times a day, maximum dose 1 g po TID beginning Day -3 until Day 35
  Arms: Double Umbilical Cord Blood Transplant

SUMMARY:
Hematopoietic cell transplants (HCT)are one treatment option for people with leukemia or lymphoma. Family members,unrelated donors or banked umbilical cordblood units with similar tissue type can be used for HCT. This study will compare the effectiveness of two new types of bone marrow transplants in people with leukemia or lymphoma: one that uses bone marrow donated from family members with only partially matched bone marrow; and, one that uses two partially matched cord blood units.

DETAILED DESCRIPTION:
Reduced intensity conditioning (RIC) blood or marrow transplantation (BMT) has allowed older and less clinically fit patients to receive potentially curative treatment with allogeneic HCT for high risk or advanced hematological malignancies. Patients lacking an HLA-matched sibling may receive a graft from a suitably HLA-matched unrelated donor. However, up to a third of patients will not have an HLA-matched sibling or a suitably matched adult unrelated donor (i.e., no more than a mismatch at a single locus). Even when a suitably matched unrelated donor is identified, data from the National Marrow Donor Program (NMDP) indicate that a median of four months is required to complete searches that result in transplantation; thus, some number of patients succumb to their disease while awaiting identification and evaluation of a suitably matched adult unrelated donor.

Single or dual center studies have shown that partially HLA-mismatched related bone marrow (haplo-BM) and unrelated double umbilical cord blood (dUCB) are valuable sources of donor cells for RIC HCT, thus extending this treatment modality to patients who lack other donors. In order to study the reproducibility, and thus, the wider applicability of these two alternative donor strategies, The Blood and Marrow Transplantation Clinical Trials Network (BMT CTN) conducted two parallel multicenter prospective Phase II clinical trials. These two studies evaluated the safety and efficacy of related haplo-BM (BMT CTN 0603) and dUCB (BMT CTN 0604) transplantation after RIC. Both of these alternative donor approaches produced early results similar to that reported with unrelated donor, and even HLA-matched sibling, HCT. These data demonstrate not only the efficacy of both of these approaches, but also that both can be safely exported from the single center setting. Both haplo-BM and dUCB grafts can be obtained rapidly for greater than 90% of patients lacking an HLA-matched donor. This study will test the hypothesis that progression free survival at two years after RIC haplo-BM transplantation is similar to the progression free survival after RIC dUCB transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 70 years old
* Patients must have available both: a)One or more potential related mismatched donors (biologic parent(s) or siblings (full or half) or children). At least low resolution DNA based human leukocyte antigen (HLA) typing at HLA-A, -B, and -DRB1 for potential haploidentical sibling donors is required. b)At least two potential umbilical cord blood units identified. Each unit must have a minimum of 1.5 x 10^7/kg pre-cryopreserved total nucleated cell dose. For non-red blood cell depleted units, the minimum pre-cryopreserved total nucleated cell dose of each unit must be at least 2.0 x 10^7/kg. Units must be HLA matched at a minimum of 4/6 to the recipient at HLA-A, HLA-B (at low resolution using DNA based typing) and HLA-DRB1 (at high resolution using DNA based typing). Confirmatory typing is not required for randomization.
* Acute Lymphoblastic Leukemia (ALL) in first complete remission (CR1) that is NOT considered favorable-risk as defined by the presence of at least one of the following: Adverse cytogenetics such as t(9;22), t(1;19), t(4;11), other Mixed Lineage Leukemia (MLL) rearrangements; White blood cell counts of greater than 30,000/mcL (B-ALL) or greater than 100,000/mcL (T-ALL)at diagnosis; Recipient age older than 30 years at diagnosis; Time to CR greater than 4 weeks
* Acute Myelogeneous Leukemia (AML) in CR1 that is NOT considered as favorable-risk. Favorable risk is defined as having one of the following: t(8.21) without CKIT mutation, inv(16) without CKIT mutation or t(16;16), normal karyotype with mutated NPM1 and not FLT-ITD, normal karyotype with double mutated CEBPA, Acute promyelocytic leukemia (APL) in first molecular remission at end of consolidation
* Acute Leukemias in 2nd or subsequent CR
* Biphenotypic/Undifferentiated/Prolymphocytic Leukemias in first or subsequent CR, adult T-cell leukemia/lymphoma in first or subsequent CR
* Burkitt's lymphoma: second or subsequent CR
* Lymphoma fulfilling the following criteria: Chemotherapy-sensitive (at least stable disease lymphomas that have failed at least 1 prior regimen of multi-agent chemotherapy and are INELIGIBLE for an autologous transplant. Patients with chronic lymphocytic leukemia (CLL) are not eligible regardless of disease status.
* Performance status: Karnofsky score greater than or equal to 70%.

Additional Patient Inclusion Criteria for Conditioning:

* Patients with Adequate Physical Function as Measured by: a. Cardiac: Left ventricular ejection fraction at rest must be greater than or equal to 40%, or shortening fraction less than 25%; b. Hepatic: Bilirubin less than or equal to 2.5 mg/dL, except for patients with Gilbert's syndrome or hemolysis. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and Alkaline Phosphatase less than 5 x upper limit of normal; c. Renal: Serum creatinine within normal range, or if serum creatinine outside normal range, then renal function (measured or estimated creatinine clearance or GFR)greater than 40 mL/min/1.73m^; d. Pulmonary: Diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin), forced expiratory volume in one second (FEV1), and forced vital capacity (FVC) greater than 50% predicted;
* Additional Patient Inclusion Criteria for Patients Assigned to Haploidentical BM Arm: Patients must be HLA typed at high resolution using DNA based typing at the following HLA-loci: HLA-A, -B, -C and DRB1 and have available a related haploidentical BM donor with 2, 3, or 4 HLA-mismatches. A unidirectional mismatch in either the graft versus host or host versus graft direction is considered a mismatch. The donor and recipient must be HLA identical for at least one antigen (using high resolution DNA based typing) at the following genetic loci: HLA-A, HLA-B, HLA-C, and HLA-DRB1. Fulfillment of this criterion shall be considered sufficient evidence that the donor and recipient share one HLA haplotype, and typing of additional family members is not required.
* Additional Patient Inclusion Criteria for Patients Assigned to Double Umbilical Cord Blood Arm:

  1. Patients must have available two UCB units fulfilling the following criteria:

     1. Each unit must have a minimum of 1.5 x 10^7/kg pre-cryopreserved total nucleated cell dose. For non-red blood cell depleted units, the minimum pre-cryopreserved total nucleated cell dose of each unit must be at least 2.0 x10^7/kg.
     2. Units must be HLA matched at a minimum of 4/6 to the recipient at HLA -A, HLA-B (at low resolution using DNA based typing), and HLA -DRB1 (at high resolution using DNA based typing).
     3. Additional graft selection criteria specified in section 2.5
  2. Patients must have received at least one cycle of the cytotoxic chemotherapy regimens (or regimen of similar intensity) listed in Appendix D within 3 months of enrollment (measured from the start date of chemotherapy) OR have had an autologous transplant within 24 months of enrollment OR receive 300 cGy as part of the preparative regimen

Exclusion Criteria:

* Patients with suitably matched related or unrelated donor, as defined per institutional practice.
* Recipients of prior autologous hematopoietic stem cell transplantation are ineligible if disease recurrence occurred less than 6 months from their autologous stem cell transplant.
* Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings).
* Prior allogeneic HCT.
* Patients with history of primary idiopathic myelofibrosis or any severe marrow fibrosis.
* Planned use of prophylactic donor lymphocyte infusion (DLI) therapy.
* Anti-donor HLA antibodies.

Additional exclusion criteria:

* Pregnancy or breast-feeding.
* Evidence of HIV infection or known HIV positive serology.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, MS, Study Director — Center for International Blood and Marrow Transplant Research (CIBMTR), Medical College of Wisconsin
Locations (39):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Cancer Center, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of California at Los Angeles, Los Angeles, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - BMT Program at Northside Hospital, Atlanta, Georgia
  - University of Kansas Hospital, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - DFCI Massachustts General Hospital, Boston, Massachusetts
  - DFCI Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute/BMT, Detroit, Michigan
  - Univeristy of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Roswell Park Cancer Center, Buffalo, New York
  - Mt. Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Jewish Hospital BMT Program, Cincinnati, Ohio
  - University Hospitals of Cleveland, Case Western, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State / Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Penn State College of Medicine - The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Univesity of Texas, MD Anderson CRC, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Eapen M, O'Donnell P, Brunstein CG, Wu J, Barowski K, Mendizabal A, Fuchs EJ. Mismatched related and unrelated donors for allogeneic hematopoietic cell transplantation for adults with hematologic malignancies. Biol Blood Marrow Transplant. 2014 Oct;20(10):1485-92. doi: 10.1016/j.bbmt.2014.05.015. Epub 2014 May 23. PMID 24862638
- [Background] Roth JA, Bensink ME, O'Donnell PV, Fuchs EJ, Eapen M, Ramsey SD. Design of a cost-effectiveness analysis alongside a randomized trial of transplantation using umbilical cord blood versus HLA-haploidentical related bone marrow in advanced hematologic cancer. J Comp Eff Res. 2014 Mar;3(2):135-44. doi: 10.2217/cer.13.95. PMID 24645687
- [Derived] Zhang P, Logan B, Martens MJ. Covariate-Adjusted Group Sequential Comparisons of Survival Probabilities. Stat Med. 2025 Dec;44(28-30):e70339. doi: 10.1002/sim.70339. PMID 41350757
- [Derived] Ramsey SD, Bansal A, Li L, O'Donnell PV, Fuchs EJ, Brunstein CG, Eapen M, Thao V, Roth JA, Steuten LMG. Cost-Effectiveness of Unrelated Umbilical Cord Blood Transplantation versus HLA-Haploidentical Related Bone Marrow Transplantation: Evidence from BMT CTN 1101. Transplant Cell Ther. 2023 Jul;29(7):464.e1-464.e8. doi: 10.1016/j.jtct.2023.04.017. Epub 2023 Apr 27. PMID 37120135
- [Derived] El Jurdi N, Martens MJ, Brunstein CG, O'Donnell P, Lee SJ, D'Souza A, Logan B, Hong S, Singh AK, Sandhu K, Shapiro RM, Horowitz MM, Hamilton BK. Health-Related Quality of Life in Double Umbilical Cord Blood versus Haploidentical Marrow Transplantation: A Quality of Life Analysis Report of BMT CTN 1101. Transplant Cell Ther. 2023 Jul;29(7):467.e1-467.e5. doi: 10.1016/j.jtct.2023.04.009. Epub 2023 Apr 22. PMID 37088401
- [Derived] Brunstein CG, DeFor TE, Fuchs EJ, Karanes C, McGuirk JP, Rezvani AR, Eapen M, O'Donnell PV, Weisdorf DJ; Blood and Marrow Transplant Clinical Trials Network. Engraftment of Double Cord Blood Transplantation after Nonmyeloablative Conditioning with Escalated Total Body Irradiation Dosing to Facilitate Engraftment in Immunocompetent Patients. Transplant Cell Ther. 2021 Oct;27(10):879.e1-879.e3. doi: 10.1016/j.jtct.2021.07.006. Epub 2021 Jul 15. PMID 34273598
- [Derived] Fuchs EJ, O'Donnell PV, Eapen M, Logan B, Antin JH, Dawson P, Devine S, Horowitz MM, Horwitz ME, Karanes C, Leifer E, Magenau JM, McGuirk JP, Morris LE, Rezvani AR, Jones RJ, Brunstein CG. Double unrelated umbilical cord blood vs HLA-haploidentical bone marrow transplantation: the BMT CTN 1101 trial. Blood. 2021 Jan 21;137(3):420-428. doi: 10.1182/blood.2020007535. PMID 33475736

RESULTS

PARTICIPANT FLOW:
Groups:
- dUCB: Participants will receive double unrelated cord blood transplant using a reduced intensity conditioning regimen.
  Double unrelated cord blood Transplant: The conditioning regimen consists of:
  * Fludarabine 40 mg/m2 IV Days -6, -5, -4, -3, -2
  * Cyclophosphamide 50 mg/kg IV Day -6
  * Total Body Irradiation (TBI): - 200 cGy Day -1 for patients who have received cytotoxic chemotherapy within the last 3 months or an autologous transplant within 24 months of enrollment; - 300 cGY Day -1 for patients who have not received cytotoxic chemotherapy within 3 months of enrollment or an autologous transplant within 24 months of enrollment
  * Day 0 will be the day of the double UCB transplant
  The GVHD prophylaxis regimen consists of:
  * Cyclosporine beginning Day -3 with dose adjusted to maintain a trough level of 200-400 ng/mL. Tacrolimus (trough level of 5-15 ng/mL) may be substituted for cyclosporine if the patient is intolerant of cyclosporine or per institutional practice.
  * Mycophenolate mofetil (MMF) 15 mg/kg po TID, maximum dose 1 g po TID beginning Day-3 until Day 35
  Supportive care includes:
  - Filgrastim (G-CSF) 5 mcg/kg/day beginning Day 1 until ANC >1500/mm3 for 3 consecutive measurements on at least two different days
- Haplo-BM: Participants will receive haploidentical bone marrow transplant using a reduced intensity conditioning regimen.
  Haploidentical Bone Marrow Transplant: The conditioning regimen consists of:
  * Fludarabine (Flu)30 mg/m2 IV Days -6, -5, -4, -3, -2
  * Cyclophosphamide (Cy) 14.5 mg/kg IV Days -6, -5
  * Total body irradiation (TBI) 200cGy Day -1
  * Day 0 will be the day of infusion of non-T-cell depleted bone marrow
  The GVHD prophylaxis regimen consists of:
  * Cy 50 mg/kg IV Days 3, 4
  * Tacrolimus (IV or PO) beginning Day 5 with dose adjusted to maintain a trough level of 5-15 ng/mL. Cyclosporine (trough level of 200-400 ng/mL) may be substituted for tacrolimus if the patient is intolerant of tacrolimus or per institutional practice.
  * Mycophenolate mofetil (MMF) 15 mg/kg po three times a day, maximum dose 1 g po TID beginning Day 5 until Day 35
  Supportive care includes:
  - Filgrastim (G-CSF) 5 mcg/kg/day beginning Day 5 until ANC >1500/mm3 for 3 consecutive measurements on at least two different days
Period: Overall Study
Arm/Group | dUCB | Haplo-BM
Started | 186 | 182
Completed | 172 | 153
Not Completed | 14 | 29
Not completed — Death | 7 | 10
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 11
Not completed — Transplanted off protocol | 2 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for all enrolled participants by treatment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | dUCB | Haplo-BM | Total
Number analyzed (Participants) | 186 | 182 | 368
Age, Continuous [Median (Full Range); unit: years]
  Median (Range) | 58.2 [19.7 to 70.5] | 59.9 [19.7 to 70.6] | 58.8 [19.7 to 70.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 76 | 165
  Male | 97 | 106 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 21 | 43
  Not Hispanic or Latino | 164 | 159 | 323
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 9 | 15 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 27 | 34 | 61
  White | 145 | 126 | 271
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Karnofsky Performance Score [Count of Participants; unit: Participants] — KPS describes patient-perceived global quality of life and functioning on a scale of 0-100.
  100: No evidence of disease; 90: Normal activity. Minor signs or symptoms of disease; 80: Normal activity with effort. Some signs or symptoms of disease; 70: Cares for self. Unable to continue normal activity; 60: Needs occasional assistance, but cares for most personal needs; 50: Needs considerable assistance and medical care; 40: Disabled. Needs special care and assistance; 30: Severely disabled. Hospital admission indicated; 20: Very sick. Active supportive therapy needed; 10: Moribund; 0: Dead
  Participants
    >=90 | 126 | 111 | 237
    <90 | 59 | 71 | 130
    Missing | 1 | 0 | 1
Primary Diagnosis [Count of Participants; unit: Participants]
  Acute Lymphoblastic Leukemia | 31 | 32 | 63
  Acute Myelogeneous Leukemia | 98 | 98 | 196
  Biphenotypic/Undifferentiated/Prolymphocytic Leukemia | 1 | 5 | 6
  Hodgkin's Lymphoma | 10 | 8 | 18
  Large Cell Lymphoma | 21 | 19 | 40
  Follicular Non-Hodgkin's Lymphoma | 7 | 5 | 12
  T-cell Leukemia/Lymphoma | 4 | 3 | 7
  Mantle Cell Lymphoma | 6 | 5 | 11
  Other Lymphoma | 8 | 7 | 15
Disease Risk for Leukemia Patients (N=272) [Count of Participants; unit: Participants] — Remission is defined as < 5% blasts with no morphological characteristics of acute leukemia (e.g., Auer Rods) in a bone marrow with > 20% cellularity, peripheral blood counts showing ANC >1000/µl, including patients in CRp. Population: Disease risk is assessed in enrolled Leukemia patients.
  Participants
    number analyzed (Participants) | 134 | 138 | 272
    First Complete Remission | 99 | 117 | 216
    Second Complete Remission | 35 | 20 | 55
    Third or More | 0 | 1 | 1
Disease Risk for Lymphoma Patients (N=96) [Count of Participants; unit: Participants] — Complete Response is defined as disappearance of all evidence of disease. Partial Response is defined as regression of measurable disease and no new sites. Population: Disease risk is assessed in enrolled Lymphoma patients.
  Participants
    number analyzed (Participants) | 52 | 44 | 96
    Complete Response | 20 | 14 | 34
    Partial Response | 25 | 25 | 50
    Follicular or Non-Hodgkin's | 7 | 5 | 12
Cytogenetics for Leukemia [Count of Participants; unit: Participants] — For Adult acute myeloid leukemia (AML), Favorable: t(15:17), inv(16), del(16q), t(16:16), [t(8:21) without del(9q) or complex]; Intermediate: normal karyotype, +6, +8, -Y, del(12p), 11q23, t(9:11); Poor: complex karyotype, -5/del(5q), -7/del(7q), abn(3q, 9q, 11q, 21q, 17p), t(6:9), t(9:22).
  For Acute lymphocytic leukemia (ALL), Poor: Ph+/t(9:22), t(4:11), 11q23, MLL, hypodiploid, t(8:14), complex.
  For Chronic lymphocytic leukemia (CLL), Intermediate: other; Poor: 17p-, 11q-, complex (>= 5). Population: Cytogenetics data on leukemia participants were retrieved from CIBMTR. Data is only measured in enrolled Leukemia patients.
  Participants
    number analyzed (Participants) | 134 | 138 | 272
    Favorable | 17 | 20 | 37
    Intermediate | 61 | 56 | 117
    Poor | 43 | 45 | 88
    Not Available | 13 | 17 | 30
HLA Matching Score for Haploidentical Donor at Randomization [Count of Participants; unit: Participants] — HLA Match Score includes genetic matching information at HLA-A, -B, and -DRB1 loci or HLA-A, -B, -C, and -DRB1 loci. Matching at all HLA-A, -B, and -DRB1 loci is designated as 6/6 HLA matching. A 4/6 HLA match includes mismatches at any two loci. Matching at all HLA-A, -B, -C, and -DRB1 loci is designated as 8/8 HLA matching. A 6/8 HLA match includes mismatches at any two loci.
  Note: *Not required if potential haplo-donor is a biological parent or child
  Participants
    3/6 | 46 | 39 | 85
    4/6 | 22 | 16 | 38
    4/8 | 0 | 1 | 1
    5/8 | 1 | 0 | 1
    6/8 | 1 | 1 | 2
    Not Required* | 116 | 125 | 241
HLA Matching Score for Cord Blood Unit 1 at Enrollment [Count of Participants; unit: Participants] — Matching at all HLA-A, -B, and -DRB1 loci is designated as 6/6 HLA matching. A 4/6 HLA match includes mismatches at any two loci.
  Participants
    4/6 | 83 | 82 | 165
    5/6 | 73 | 75 | 148
    6/6 | 30 | 25 | 55
HLA Matching Score for Cord Blood Unit 2 at Enrollment [Count of Participants; unit: Participants] — Matching at all HLA-A, -B, and -DRB1 loci is designated as 6/6 HLA matching. A 4/6 HLA match includes mismatches at any two loci.
  Participants
    4/6 | 99 | 99 | 198
    5/6 | 66 | 64 | 130
    6/6 | 21 | 19 | 40
Pre-cryopreservation total nucleated cell count [Median (Full Range); unit: cells x 10^7/kg] — Population: Statistics is summarized on available data.
  cells x 10^7/kg
    number analyzed (Participants) | 166 | 11 | 177
    (all) | 5.13 [1.68 to 27.46] | 5.59 [3.00 to 8.72] | 5.15 [1.68 to 27.46]
Post-thaw total nucleated cell count [Median (Full Range); unit: cells x 10^7/kg] — Population: Statistics is summarized on available data.
  cells x 10^7/kg
    number analyzed (Participants) | 72 | 5 | 77
    (all) | 4.32 [0.04 to 9.23] | 3.12 [2.80 to 7.51] | 4.32 [0.04 to 9.23]
Total nucleated cell count at infusion [Median (Full Range); unit: cells x 10^7/kg] — Population: Statistics is summarized on available data.
  cells x 10^7/kg
    number analyzed (Participants) | 167 | 121 | 288
    (all) | 2.95 [0.01 to 84.09] | 26.82 [0.19 to 73.50] | 4.46 [0.01 to 84.09]
Pre-cryopreservation CD34+ cell count [Median (Full Range); unit: cells x 10^6/kg] — Population: Statistics is summarized on available data.
  cells x 10^6/kg
    number analyzed (Participants) | 157 | 11 | 168
    (all) | 0.23 [0.03 to 1.22] | 0.21 [0.11 to 0.29] | 0.22 [0.03 to 1.22]
Post-thaw CD34+ cell count [Median (Full Range); unit: cells x 10^6/kg] — Population: Statistics is summarized on available data.
  cells x 10^6/kg
    number analyzed (Participants) | 66 | 5 | 71
    (all) | 0.20 [0.00 to 0.76] | 0.17 [0.13 to 0.34] | 0.20 [0.00 to 0.76]
CD34+ cell count at infusion [Median (Full Range); unit: cells x 10^6/kg] — Population: Statistics is summarized on available data.
  cells x 10^6/kg
    number analyzed (Participants) | 155 | 73 | 228
    (all) | 0.13 [0.00 to 1.20] | 2.87 [0.03 to 235.14] | 0.20 [0.00 to 235.14]
Pre-cryopreservation CD3+ cell count [Median (Full Range); unit: cells x 10^6/kg] — Population: Statistics is summarized on available data.
  cells x 10^6/kg
    number analyzed (Participants) | 7 | 1 | 8
    (all) | 7.79 [0.00 to 15.82] | 0.00 [0.00 to 0.00] | 7.38 [0.00 to 15.82]
Post-thaw CD3+ cell count [Median (Full Range); unit: cells x 10^6/kg] — Population: Statistics is summarized on available data.
  cells x 10^6/kg
    number analyzed (Participants) | 49 | 2 | 51
    (all) | 6.97 [0.03 to 29.03] | 7.47 [5.21 to 9.73] | 6.97 [0.03 to 29.03]
CD3+ cell count at infusion [Median (Full Range); unit: cells x 10^6/kg] — Population: Statistics is summarized on available data.
  cells x 10^6/kg
    number analyzed (Participants) | 111 | 71 | 182
    (all) | 5.50 [0.00 to 165.88] | 29.66 [0.48 to 548.87] | 8.05 [0.00 to 548.87]
HCT-comorbidity index (CI) [Count of Participants; unit: Participants] — The HCT-CI was developed to identify comorbidities relevant to transplant and act as a tool for risk assessment and before allogeneic hematopoietic stem cell transplantation. Patients with no comorbidities are assigned a score of zero. Arrhythmia, cardiac, bowel, diabetes, cerebrovascular, psychological, mild chronic hepatitis, obesity, infection are assigned a score of 1. Rheumatoid arthritis, peptic ulcer, renal moderate/severe, pulmonary moderate, are assigned a score of 2. Solid tumor, heart valve disease, pulmonary sever, hepatic moderate/severe are assigned a score of 3. Population: HCT-CI was only measured in the transplanted participants. The total number of participants is different from the overall number of enrolled participants as 11 participants from dUCB arm and 15 participants from Haplo-BM arm were not transplanted.
  Participants
    number analyzed (Participants) | 175 | 167 | 342
    >=3 | 71 | 68 | 139
    2 | 26 | 23 | 49
    1 | 26 | 23 | 49
    0 | 52 | 53 | 105
CMV Status at Transplant [Count of Participants; unit: Participants] — Cytomegalovirus (CMV) status Population: CMV status was only measured in the transplanted participants. The total number of participants is different from the overall number of enrolled participants as 11 participants from dUCB arm and 15 participants from Haplo-BM arm were not transplanted.
  Participants
    number analyzed (Participants) | 175 | 167 | 342
    Positive | 98 | 99 | 197
    Negative | 76 | 68 | 144
    Missing | 1 | 0 | 1
Time from Diagnosis to Transplant [Median (Full Range); unit: day] — Population: Time to transplant was only calculated in the transplanted participants. The total number of participants is different from the overall number of enrolled participants as 11 participants from dUCB arm and 15 participants from Haplo-BM arm were not transplanted.
  day
    number analyzed (Participants) | 175 | 167 | 342
    (all) | 283 [53 to 7383] | 219 [50 to 7952] | 233 [50 to 7952]
Prior Autologous Transplant [Count of Participants; unit: Participants]
  Prior Autologous Transplant | 16 | 16 | 32
  No Prior Autologous Transplant | 170 | 166 | 336
Number of Regimens Prior to Transplant [Count of Participants; unit: Participants] — Population: Number of regimens prior to transplant was only counted in the transplanted participants. The total number of participants is different from the overall number of enrolled participants as 11 participants from dUCB arm and 15 participants from Haplo-BM arm were not transplanted.
  Participants
    number analyzed (Participants) | 175 | 167 | 342
    5 | 4 | 7 | 11
    4 | 6 | 6 | 12
    3 | 14 | 8 | 22
    2 | 8 | 10 | 18
    1 | 17 | 10 | 27
    0 | 2 | 0 | 2
    Unknown | 124 | 126 | 250
Disease Risk Index [Count of Participants; unit: Participants] — The disease risk index was computed based on participant's primary diagnosis, disease risk and cytogenetic data.
  Participants
    Low | 23 | 14 | 37
    Intermediate | 119 | 120 | 239
    High | 35 | 37 | 72
    Not Available | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS)
Description: The primary endpoint is PFS at 2 years post-randomization. Death or disease relapse/progression will be considered as events. The time to event is defined as the time interval from randomization to relapse/progression, to death or to last follow-up, whichever comes first. Relapse is defined by either morphological or cytogenetic evidence of acute leukemia consistent with pre-transplant features, or radiologic evidence of progressive lymphoma. Minimal residual disease will not be considered evidence of relapse, however, minimal residual disease that progresses will be considered as relapse and the date of relapse will be the date of detection of minimal residual disease that prompted an intervention by the treating physician. Finally, institution of any therapy to treat persistent, progressive or relapsed disease, including withdrawal of immunosuppressive therapy or DLI, will be considered evidence of relapse/progression regardless of whether the criteria described above are met.
Time Frame: Year 2
Population: The primary endpoint analysis is performed using the intent-to-treat principle so that all randomized patients are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 186 | 182
percentage of participants | 35.0 [28.0 to 42.1] | 41.1 [33.6 to 48.4]
Statistical Analysis 1: Comparison: dUCB vs Haplo-BM; The primary null hypothesis of the study is that there is no difference between the 2 year PFS probabilities for dUCB vs. haplo-BM; Test type: Superiority; p = 0.4092, Z-test to compare the Kaplan-Meier Est. — Statistical significance was determined using a pre-specified threshold of 0.05. Final p-value is adjusted for the interim looks per study design; Difference in Kaplan-Meier estimates = 6.1, 95% CI 2-sided [-5.2 to 17.4]
Statistical Analysis 2: Comparison: dUCB vs Haplo-BM; The null hypothesis of the study is that there is no difference between the 2 year PFS probabilities for dUCB vs. haplo-BM after adjustment for age, performance score, and disease type; Test type: Superiority; p = 0.060, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.99 to 1.70]

2. Secondary Outcome: Percentage of Participants With PFS by Treatment Arms in Subgroups
Description: Participants' primary diagnosis was categorized into two large groups: leukemia versus lymphoma. Age was dichotomized into two large groups: age <= 59 versus age > 59. The Kaplan-Meier estimate for PFS at 2 years post-randomization are provided for each subgroup.
Time Frame: Year 2
Population: The randomized participants are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 186 | 182
percentage of participants
  By Primary Disease of Leukemia: number analyzed (Participants) | 134 | 138
  By Primary Disease of Leukemia | 34.8 [26.6 to 43.1] | 41.7 [33.0 to 50.1]
  By Primary Disease of Lymphoma: number analyzed (Participants) | 52 | 44
  By Primary Disease of Lymphoma | 35.6 [22.7 to 48.6] | 39.3 [24.7 to 53.5]
  By Age Group <= 59 years: number analyzed (Participants) | 101 | 86
  By Age Group <= 59 years | 37.9 [28.2 to 47.5] | 39.6 [28.8 to 50.2]
  By Age Group > 59 years: number analyzed (Participants) | 85 | 96
  By Age Group > 59 years | 31.6 [21.8 to 41.9] | 42.4 [32.1 to 52.3]

3. Secondary Outcome: Percentage of Participants With Neutrophil Recovery
Description: Neutrophil recovery is defined as achieving an absolute neutrophil count greater than or equal to 500/mm^3 for three consecutive measurements on three different days. The first of the three days will be designated the day of neutrophil recovery.
Time Frame: Day 56
Population: The transplanted participants are included in the analysis. A total of 26 patients (11 on the dUCB arm and 15 on the Haplo-BM arm) who did not proceed to the study transplant are excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 175 | 167
percentage of participants | 94.9 [90.2 to 97.4] | 98.8 [94.3 to 99.8]
Statistical Analysis 1: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the neutrophil engraftment post-transplantation for dUCB vs. haplo-BM; Test type: Superiority; p = 0.046, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05; Estimate cumulative incidence functions from competing risks data and test equality of 2 trt grps. Death before neutrophil recovery is competing risk

4. Secondary Outcome: Percentage of Participants With Platelet Recovery
Description: Platelet recovery is defined by two different metrics as the first day of a sustained platelet count greater than 20,000/mm^3 or greater than 50,000/mm^3 with no platelet transfusions in the preceding seven days. The first day of the sustained platelet count will be designated the day of platelet engraftment.
Time Frame: Day 100
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 175 | 167
percentage of participants
  Platelet recovery to 20K | 86.9 [80.8 to 91.2] | 91.6 [86.1 to 95.0]
  Platelet recovery to 50K | 78.3 [71.4 to 83.7] | 84.4 [77.9 to 89.1]
Statistical Analysis 1: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the platelet engraftment to 20k post-transplantation for dUCB vs. haplo-BM; Test type: Superiority; p = 0.160, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05; Estimate cumulative incidence functions from competing risks data and test equality of 2 trt grps. Death before Platelet recovery is competing risk
Statistical Analysis 2: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the platelet engraftment to 50k post-transplantation for dUCB vs. haplo-BM; Test type: Superiority; p = 0.146, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Participants With Primary Graft Failure
Description: Primary graft failure is defined as less than 5% donor chimerism on all measurements up to and including Day 56.
Time Frame: Day 56
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 175 | 167
Participants | 13 | 10

6. Secondary Outcome: Percentage of Participants With Secondary Graft Failure
Description: Secondary graft failure is defined as initial donor chimerism ≥ 5% declining to < 5% on subsequent measurements with time to secondary graft failure beginning at the first day of primary engraftment.
Time Frame: Year 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 175 | 167
percentage of participants | 2.6 [0.9 to 6.1] | 3.4 [1.3 to 7.2]
Statistical Analysis 1: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the secondary graft failure probabilities post-transplantation for dUCB vs. haplo-BM; Test type: Superiority; p = 0.693, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05; Estimate cumulative incidence functions from competing risks data and test equality of 2 trt grps. Death before 2nd graft failure is competing risk

7. Secondary Outcome: Percentage of Participants With Acute Graft-versus-Host Disease (aGVHD)
Description: The cumulative incidences of grade II - IV and III - IV acute aGVHD will be determined.
Time Frame: Day 180
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 175 | 167
percentage of participants
  grade II - IV | 34.9 [27.9 to 42.0] | 28.1 [21.5 to 35.1]
  grade III - IV | 8.6 [5.0 to 13.3] | 7.2 [3.9 to 11.8]
Statistical Analysis 1: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the aGVHD grade II - IV probabilities post-transplantation for dUCB vs. haplo-BM; Test type: Superiority; p = 0.142, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05; Estimate cumulative incidence functions from competing risks data and test equality of 2 trt grps. Death prior to aGVHD is competing risk
Statistical Analysis 2: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the aGVHD grade III - IV probabilities post-transplantation for dUCB vs. haplo-BM; Test type: Superiority; p = 0.604, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 7, analysis 1]

8. Secondary Outcome: Percentage of Participants With Chronic Graft-versus-Host Disease (cGHVD)
Description: The cumulative incidence of cGVHD from the time of transplant will be determined. Data were collected directly from providers and chart review according to the recommendations of the NIH Consensus Conference.
Time Frame: Year 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 175 | 167
percentage of participants | 22.0 [16.1 to 28.5] | 26.2 [19.7 to 33.2]
Statistical Analysis 1: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the cGVHD probabilities post-transplantation for dUCB vs. haplo-BM; Test type: Superiority; p = 0.361, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05; Estimate cumulative incidence functions from competing risks data and test equality of 2 trt grps. Death before cGVHD is competing risk

9. Secondary Outcome: Percentage of Participants With Overall Survival
Description: Overall survival is defined as the time interval between date of randomization and death from any cause or for surviving patients, to last follow-up. The time interval between date of transplant and death from any cause or for surviving patients, to last follow-up are also analyzed.
Time Frame: Year 2
Population: The randomized or transplanted participants are included in the analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 186 | 182
percentage of participants
  OS post-randomization | 45.7 [38.1 to 53.0] | 57.0 [49.1 to 64.2]
  OS post-transplant: number analyzed (Participants) | 175 | 167
  OS post-transplant | 46.8 [38.9 to 54.2] | 59.4 [51.2 to 66.7]
Statistical Analysis 1: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the OS probabilities at year 2 post-randomization for dUCB vs. haplo-BM; Test type: Superiority; p = 0.0373, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the OS probabilities at year 2 post-transplant for dUCB vs. haplo-BM; Test type: Superiority; p = 0.0235, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05

10. Secondary Outcome: Percentage of Participants With Treatment-related Mortality (TRM)
Description: The cumulative incidence of TRM will be estimated, event for this endpoint is death without evidence of disease progression or recurrence.
Time Frame: Day 100, Day 180, Year 1, and Year 2
Population: The randomized or transplanted participants are included in the analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 186 | 182
percentage of participants
  Day 100 Post Randomization | 5.5 [2.8 to 9.4] | 3.4 [1.4 to 6.8]
  Day 100 Post Transplant: number analyzed (Participants) | 175 | 167
  Day 100 Post Transplant | 6.9 [3.7 to 11.3] | 3.6 [1.5 to 7.2]
  Day 180 Post Randomization | 10.4 [6.5 to 15.3] | 4.5 [2.1 to 8.2]
  Day 180 Post Transplant: number analyzed (Participants) | 175 | 167
  Day 180 Post Transplant | 13.1 [8.6 to 18.6] | 4.8 [2.2 to 8.8]
  1 Year Post Randomization | 14.8 [10.1 to 20.3] | 6.7 [3.7 to 11.1]
  1 Year Post Transplant: number analyzed (Participants) | 175 | 167
  1 Year Post Transplant | 16.0 [11.0 to 21.9] | 7.9 [4.4 to 12.7]
  2 Year Post Randomization | 17.9 [12.7 to 23.9] | 10.5 [6.5 to 15.7]
  2 Year Post Transplant: number analyzed (Participants) | 175 | 167
  2 Year Post Transplant | 18.6 [13.1 to 24.8] | 10.7 [6.5 to 16.1]
Statistical Analysis 1: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the TRM probabilities post-randomization for dUCB vs. haplo-BM; Test type: Superiority; p = 0.039, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05; Estimate cumulative incidence functions from competing risks data and test equality across the two treatment groups
Statistical Analysis 2: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the TRM probabilities post-transplantation for dUCB vs. haplo-BM; Test type: Superiority; p = 0.030, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05; Estimate cumulative incidence functions from competing risks data and test equality across the two treatment groups

11. Secondary Outcome: Percentage of Participants With Relapse/Progression
Description: Incidence of relapse/progression will be estimated using cumulative incidence function, treating death in remission as a competing risk. Relapse is defined by either morphological or cytogenetic evidence of acute leukemia consistent with pre-transplant features, or radiologic evidence of progressive lymphoma. When in doubt, the diagnosis of recurrent or progressive lymphoma should be documented by tissue biopsy. Minimal residual disease will not be considered evidence of relapse, however, minimal residual disease that progresses will be considered as relapse and the date of relapse will be the date of detection of minimal residual disease that prompted an intervention by the treating physician. Finally, institution of any therapy to treat persistent, progressive or relapsed disease, including withdrawal of immunosuppressive therapy or DLI, will be considered evidence of relapse/progression regardless of whether the criteria described above are met.
Time Frame: Year 1, year 2
Population: The randomized or transplanted participants are included in the analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 186 | 182
percentage of participants
  1 Year Post Randomization | 41.1 [33.9 to 48.1] | 37.6 [30.5 to 44.7]
  1 Year Post Transplant: number analyzed (Participants) | 175 | 167
  1 Year Post Transplant | 38.7 [31.4 to 46.0] | 35.1 [27.8 to 42.5]
  2 Year Post Randomization | 47.1 [39.6 to 54.2] | 48.4 [40.7 to 55.7]
  2 Year Post Transplant: number analyzed (Participants) | 175 | 167
  2 Year Post Transplant | 43.5 [35.8 to 50.9] | 45.8 [37.7 to 53.5]
Statistical Analysis 1: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the relapse/progression probabilities post-randomization for dUCB vs. haplo-BM; Test type: Superiority; p = 0.968, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05; Estimate cumulative incidence functions from competing risks data and test equality of 2 trt grps. Death prior to relapse is competing risk
Statistical Analysis 2: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the relapse/progression probabilities post- transplantation for dUCB vs. haplo-BM; Test type: Superiority; p = 0.907, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 11, analysis 1]

12. Secondary Outcome: Toxicities
Description: They are all Grade ≥ 3 toxicities based on NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.
Time Frame: Day 28, Day 56, Day 180, 1 year, and 2 years
Population: as for outcome 3
Measure: Number; unit: Toxicities
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 175 | 167
Toxicities
  Toxicities Reported at Day 0-28 : Infusion Toxicities | 19 | 7
  Toxicities Reported at Day 0-28 : Oral Mucositis | 2 | 2
  Toxicities Reported at Day 0-28 : Cystitis Noninfective | 1 | 1
  Toxicities Reported at Day 0-28 : Acute Kidney Injury | 4 | 4
  Toxicities Reported at Day 0-28 : Chronic Kidney Disease | 0 | 2
  Toxicities Reported at Day 0-28 : Hemorrhage | 2 | 6
  Toxicities Reported at Day 0-28 : Hypotension | 12 | 10
  Toxicities Reported at Day 0-28 : Cardiac Arrhythmia | 6 | 6
  Toxicities Reported at Day 0-28 : Left Ventricular Systolic Dysfunction | 2 | 0
  Toxicities Reported at Day 0-28 : Somnolence | 2 | 1
  Toxicities Reported at Day 0-28 : Thrombotic Thrombocytopenic Purpura | 3 | 1
  Toxicities Reported at Day 0-28 : Capillary Leak Syndrome | 1 | 0
  Toxicities Reported at Day 0-28 : Hypoxia | 9 | 9
  Toxicities Reported at Day 0-28 : Dyspnea | 7 | 0
  Toxicities Reported at Day 0-28 : ALT | 3 | 6
  Toxicities Reported at Day 0-28 : AST | 2 | 4
  Toxicities Reported at Day 0-28 : Bilirubin | 3 | 1
  Toxicities Reported at Day 0-28 : Alkaline Phosphatase | 4 | 1
  Toxicities Reported at Day 0-28 : Abnormal Liver Symptoms | 2 | 4
  Toxicities Reported at Day 0-28 : Received Dialysis | 2 | 1
  Toxicities Reported at Day 0-28 : Seizure | 0 | 0
  Toxicities Reported at Day 29-56 : Infusion Toxicities | 0 | 0
  Toxicities Reported at Day 29-56 : Oral Mucositis | 3 | 2
  Toxicities Reported at Day 29-56 : Cystitis Noninfective | 2 | 1
  Toxicities Reported at Day 29-56 : Acute Kidney Injury | 3 | 3
  Toxicities Reported at Day 29-56 : Chronic Kidney Disease | 2 | 3
  Toxicities Reported at Day 29-56 : Hemorrhage | 2 | 4
  Toxicities Reported at Day 29-56 : Hypotension | 5 | 5
  Toxicities Reported at Day 29-56 : Cardiac Arrhythmia | 3 | 2
  Toxicities Reported at Day 29-56 : Left Ventricular Systolic Dysfunction | 2 | 1
  Toxicities Reported at Day 29-56 : Somnolence | 4 | 1
  Toxicities Reported at Day 29-56 : Thrombotic Thrombocytopenic Purpura | 6 | 1
  Toxicities Reported at Day 29-56 : Capillary Leak Syndrome | 0 | 1
  Toxicities Reported at Day 29-56 : Hypoxia | 6 | 5
  Toxicities Reported at Day 29-56 : Dyspnea | 9 | 6
  Toxicities Reported at Day 29-56 : ALT | 7 | 1
  Toxicities Reported at Day 29-56 : AST | 5 | 1
  Toxicities Reported at Day 29-56 : Bilirubin | 3 | 1
  Toxicities Reported at Day 29-56 : Alkaline Phosphatase | 2 | 0
  Toxicities Reported at Day 29-56 : Abnormal Liver Symptoms | 4 | 4
  Toxicities Reported at Day 29-56 : Received Dialysis | 3 | 2
  Toxicities Reported at Day 29-56 : Seizure | 0 | 0
  Toxicities Reported at Day 57-180 : Infusion Toxicities | 0 | 0
  Toxicities Reported at Day 57-180 : Oral Mucositis | 1 | 1
  Toxicities Reported at Day 57-180 : Cystitis Noninfective | 1 | 2
  Toxicities Reported at Day 57-180 : Acute Kidney Injury | 9 | 7
  Toxicities Reported at Day 57-180 : Chronic Kidney Disease | 1 | 4
  Toxicities Reported at Day 57-180 : Hemorrhage | 3 | 6
  Toxicities Reported at Day 57-180 : Hypotension | 12 | 10
  Toxicities Reported at Day 57-180 : Cardiac Arrhythmia | 4 | 3
  Toxicities Reported at Day 57-180 : Left Ventricular Systolic Dysfunction | 2 | 1
  Toxicities Reported at Day 57-180 : Somnolence | 5 | 2
  Toxicities Reported at Day 57-180 : Thrombotic Thrombocytopenic Purpura | 3 | 1
  Toxicities Reported at Day 57-180 : Capillary Leak Syndrome | 1 | 0
  Toxicities Reported at Day 57-180 : Hypoxia | 22 | 7
  Toxicities Reported at Day 57-180 : Dyspnea | 21 | 8
  Toxicities Reported at Day 57-180 : ALT | 6 | 4
  Toxicities Reported at Day 57-180 : AST | 8 | 5
  Toxicities Reported at Day 57-180 : Bilirubin | 8 | 3
  Toxicities Reported at Day 57-180 : Alkaline Phosphatase | 4 | 4
  Toxicities Reported at Day 57-180 : Abnormal Liver Symptoms | 6 | 5
  Toxicities Reported at Day 57-180 : Received Dialysis | 2 | 2
  Toxicities Reported at Day 57-180 : Seizure | 0 | 0
  Toxicities Reported at Day 181-365 : Infusion Toxicities | 0 | 0
  Toxicities Reported at Day 181-365 : Oral Mucositis | 2 | 0
  Toxicities Reported at Day 181-365 : Cystitis Noninfective | 2 | 1
  Toxicities Reported at Day 181-365 : Acute Kidney Injury | 4 | 6
  Toxicities Reported at Day 181-365 : Chronic Kidney Disease | 2 | 2
  Toxicities Reported at Day 181-365 : Hemorrhage | 3 | 5
  Toxicities Reported at Day 181-365 : Hypotension | 3 | 9
  Toxicities Reported at Day 181-365 : Cardiac Arrhythmia | 4 | 5
  Toxicities Reported at Day 181-365 : Left Ventricular Systolic Dysfunction | 2 | 0
  Toxicities Reported at Day 181-365 : Somnolence | 3 | 5
  Toxicities Reported at Day 181-365 : Thrombotic Thrombocytopenic Purpura | 4 | 1
  Toxicities Reported at Day 181-365 : Capillary Leak Syndrome | 0 | 1
  Toxicities Reported at Day 181-365 : Hypoxia | 8 | 10
  Toxicities Reported at Day 181-365 : Dyspnea | 10 | 11
  Toxicities Reported at Day 181-365 : ALT | 4 | 4
  Toxicities Reported at Day 181-365 : AST | 5 | 4
  Toxicities Reported at Day 181-365 : Bilirubin | 5 | 5
  Toxicities Reported at Day 181-365 : Alkaline Phosphatase | 6 | 4
  Toxicities Reported at Day 181-365 : Abnormal Liver Symptoms | 3 | 3
  Toxicities Reported at Day 181-365 : Received Dialysis | 1 | 4
  Toxicities Reported at Day 181-365 : Seizure | 0 | 2
  Toxicities Reported at Day 363-730 : Infusion Toxicities | 0 | 0
  Toxicities Reported at Day 363-730 : Oral Mucositis | 3 | 1
  Toxicities Reported at Day 363-730 : Cystitis Noninfective | 1 | 2
  Toxicities Reported at Day 363-730 : Acute Kidney Injury | 3 | 3
  Toxicities Reported at Day 363-730 : Chronic Kidney Disease | 1 | 0
  Toxicities Reported at Day 363-730 : Hemorrhage | 2 | 0
  Toxicities Reported at Day 363-730 : Hypotension | 6 | 5
  Toxicities Reported at Day 363-730 : Cardiac Arrhythmia | 0 | 2
  Toxicities Reported at Day 363-730 : Left Ventricular Systolic Dysfunction | 0 | 1
  Toxicities Reported at Day 363-730 : Somnolence | 0 | 4
  Toxicities Reported at Day 363-730 : Thrombotic Thrombocytopenic Purpura | 1 | 0
  Toxicities Reported at Day 363-730 : Capillary Leak Syndrome | 0 | 0
  Toxicities Reported at Day 363-730 : Hypoxia | 6 | 7
  Toxicities Reported at Day 363-730 : Dyspnea | 4 | 8
  Toxicities Reported at Day 363-730 : ALT | 1 | 4
  Toxicities Reported at Day 363-730 : AST | 0 | 4
  Toxicities Reported at Day 363-730 : Bilirubin | 1 | 3
  Toxicities Reported at Day 363-730 : Alkaline Phosphatase | 1 | 3
  Toxicities Reported at Day 363-730 : Abnormal Liver Symptoms | 2 | 5
  Toxicities Reported at Day 363-730 : Received Dialysis | 1 | 2
  Toxicities Reported at Day 363-730 : Seizure | 0 | 1
  Overall Toxicities Reported Day 0-730: Infusion Toxicities | 19 | 7
  Overall Toxicities Reported Day 0-730: Oral Mucositis | 9 | 6
  Overall Toxicities Reported Day 0-730: Cystitis Noninfective | 6 | 6
  Overall Toxicities Reported Day 0-730: Acute Kidney Injury | 22 | 19
  Overall Toxicities Reported Day 0-730: Chronic Kidney Disease | 5 | 9
  Overall Toxicities Reported Day 0-730: Hemorrhage | 12 | 12
  Overall Toxicities Reported Day 0-730: Hypotension | 31 | 32
  Overall Toxicities Reported Day 0-730: Cardiac Arrhythmia | 14 | 14
  Overall Toxicities Reported Day 0-730: Left Ventricular Systolic Dysfunction | 8 | 3
  Overall Toxicities Reported Day 0-730: Somnolence | 13 | 13
  Overall Toxicities Reported Day 0-730: Thrombotic Thrombocytopenic Purpura | 14 | 4
  Overall Toxicities Reported Day 0-730: Capillary Leak Syndrome | 2 | 2
  Overall Toxicities Reported Day 0-730: Hypoxia | 41 | 34
  Overall Toxicities Reported Day 0-730: Dyspnea | 38 | 35
  Overall Toxicities Reported Day 0-730: ALT | 18 | 19
  Overall Toxicities Reported Day 0-730: AST | 19 | 18
  Overall Toxicities Reported Day 0-730: Bilirubin | 18 | 13
  Overall Toxicities Reported Day 0-730: Alkaline Phosphatase | 14 | 12
  Overall Toxicities Reported Day 0-730: Abnormal Liver Symptoms | 15 | 18
  Overall Toxicities Reported Day 0-730: Received Dialysis | 8 | 9
  Overall Toxicities Reported Day 0-730: Seizure | 0 | 3

13. Secondary Outcome: Participants With Infections
Description: All Grade 2 and 3 infections will be reported. Grade 1 CMV infections through Day 56 will also be reported.
Time Frame: Up to 2 years
Population: The transplanted participants are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 175 | 167
Participants
  # Patients with Infections | 102 | 102
  Grade 1 CMV through Day 56 | 94 | 84

14. Secondary Outcome: Hospital Admission and Length of Stay
Description: Total Time Alive and Not Hospitalized within 6 Months Post Randomization
Time Frame: Month 6
Population: The randomized participants are included in the analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | dUCB | Haplo-BM
Number analyzed (Participants) | 186 | 182
Days | 127.1 (48.3) | 141.2 (42.5)
Statistical Analysis 1: Comparison: dUCB vs Haplo-BM; The null hypothesis is that there is no difference between the total duration of hospitalization within 6 months post-randomization for dUCB vs. haplo-BM; Test type: Superiority; p = 0.0003, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

ADVERSE EVENTS:
Time Frame: Adverse event reporting and monitoring were conducted throughout the study, up to 2 years.
Description: Adverse event (AE) reporting was conducted according to the BMT CTN's manual of operating procedures (MOP). Unexpected, grade 3-5 AE were reported through an expedited AE reporting system. Expected AEs were reported using National Cancer Institute (NCI)'s Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 at regular intervals and reported in the secondary outcome "Toxicities". All fatal (Grade 5) expected adverse events were reported in an expedited manner.
Arm/Group | dUCB | Haplo-BM
All-Cause Mortality (participants affected / at risk) | 97/186 | 74/182
Serious Adverse Events (participants affected / at risk) | 4/186 | 9/182
Other Adverse Events (participants affected / at risk) | 1/186 | 0/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dUCB (N=186) | Haplo-BM (N=182)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) — Cardiorespiratory
Supraventricular tachycardia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Supraventricular tachycardia
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Arterial injury
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Infusion related reaction
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Vascular access complication
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Acute myeloid leukemia
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1) — Central nervous system lesion
Syncope (Nervous system disorders) | 0 (0) | 1 (1) — Syncope
Psychiatric disorders Delirium (Psychiatric disorders) | 1 (1) | 0 (0) — Psychiatric disorders Delirium
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Respiratory failure
Embolism (Vascular disorders) | 0 (0) | 1 (1) — Embolism
Hypotension (Vascular disorders) | 0 (0) | 1 (1) — Hypotension
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dUCB (N=186) | Haplo-BM (N=182)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — MYELODYSPLASTIC SYNDROME

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT01597778/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT01597778/SAP_001.pdf
  • Informed Consent Form (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT01597778/ICF_002.pdf